CLINICAL TRIAL: NCT05136014
Title: Evaluation of the Response to Tyrosine Kinase Inhibitors in Localized Non-small Cell Lung Cancer (NSCLC) Patients With EGFR Mutation in a Patient-derived Organoid Model
Acronym: OS-TUMOVASC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Principal Investigator, SEITLINGER Joseph, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI057
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer; Lung Adenocarcinoma; EGFR Activating Mutation; KRAS Mutation-Related Tumors; Non Small Cell Lung Cancer
Keywords: tyrosine kinase inhibitors; Lung adenocarcinoma; EGFR activating mutation; KRAS Mutation-related tumors
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General cohorte: patient with non-small cell lung cancer undergoing surgical resection in the thoracic surgery department of the Nancy CHRU
  Interventions: Other: Collection of surgical waste

INTERVENTIONS:
Other: Collection of surgical waste — collection of a fragment of healthy and tumorous lung tissue taken as part of the operating theatre procedure and normally destined to be destroyed

SUMMARY:
Lung cancer is a major public health problem and remains the leading cause of cancer mortality worldwide. Moreover, in France, it is the 3rd most common cancer in terms of incidence. Its prognosis remains poor despite the emergence of new therapies, notably the Epithelial Growth Factor Receptor (EGFR) specific tyrosine kinase inhibitors which can be used in patients with adenocarcinoma presenting an activating mutation of EGFR.

In addition, a number of questions remain regarding the use of these molecules, including the possibility of combining them with other therapies such as chemotherapy or radiotherapy. In addition, the duration of treatment with tyrosine kinase inhibitors is a matter of debate, mainly in localised forms (ADAURA trial). For this reason, we have proposed tests using TKIs on an in vitro platform based on organoid formation from tumour biopsies of NSCLC patients. This model will allow to test different molecules, in particular osimertinib which is a third generation tyrosine kinase inhibitor. In this way, it will be possible to evaluate in vitro responder patients within a timeframe compatible with the timeframe proposed by the INCA (4-6 weeks).

For non-responders, it will also be possible to screen them in vitro and seek the ideal alternative therapy. This model therefore aims to develop personalised medicine in thoracic oncology and could be used as a decision aid during multidisciplinary consultation meetings.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* patient affiliated to a social security scheme
* having given their agreement to participate in the study
* with non small cell lung cancer of any stage undergoing surgical resection at the Nancy University Hospital

Exclusion Criteria:

* Refusal to participate
* Hepatitis
* HIV
* Legal guardianship
* Guardianship
* Inability to give informed information to the patient
* Pregnant women-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non small cell lung cancer of any stage undergoing surgical resection at the Nancy University Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the in vitro efficacy of osimertinib in a patient-derived organoid model alone or in combination | from day 0 to day 30
  Cell viability test

SECONDARY OUTCOMES:
Identify non-responders to osimertinib in vitro | from day 0 to day 30
  Cell viability test

CONTACTS AND LOCATIONS:
Locations (1):
- Seitlinger, Vandœuvre-lès-Nancy, Lorraine, France